CLINICAL TRIAL: NCT03359460
Title: Phase I Trial of the Combination of Ibrutinib and Lenalidomide for the Treatment of Patients With MDS Who Have Failed or Refuse Standard Therapy
Brief Title: Ibrutinib and Lenalidomide in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brian Jonas (Other)
Collaborators: Pharmacyclics LLC. (Industry); Celgene (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Brian Jonas, Principal Investigator, University of California, Davis
Organization: University of California, Davis (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1043625; UCDCC#265 (Other: UC Davis); UCDCC#265 (Other: University of California Davis Comprehensive Cancer Center); P30CA093373 (NIH); NCI-2017-01827 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Myelodysplastic Syndrome; Previously Treated Myelodysplastic Syndrome; Refractory High Risk Myelodysplastic Syndrome; Secondary Myelodysplastic Syndrome; Therapy-Related Myelodysplastic Syndrome
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — ibrutinib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (lenalidomide, ibrutinib) (Experimental): Patients receive lenalidomide PO QD on days 1-21 and ibrutinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unaccepted toxicity.
  Interventions: Drug: Ibrutinib; Drug: Lenalidomide

INTERVENTIONS:
Drug: Ibrutinib — Given PO
  Other Names: BTK Inhibitor PCI-32765; CRA-032765; Imbruvica; PCI-32765
Drug: Lenalidomide — Given PO
  Other Names: CC-5013; CC5013; CDC 501; Revlimid

SUMMARY:
This phase I trial studies the side effects and best dose of ibrutinib when giving together with lenalidomide in treating patients with myelodysplastic syndrome. Ibrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as lenalidomide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving ibrutinib and lenalidomide may work better in treating patients with myelodysplastic syndrome.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To determine the recommended Phase II dose (RP2D) for ibrutinib in combination with lenalidomide in patients with myelodysplastic syndrome (MDS).

SECONDARY OBJECTIVES:

To do an early assessment of the activity of the combination of ibrutinib and lenalidomide in patients with MDS.

TERTIARY OBJECTIVES:

To examine the pharmacodynamic and biological effects of the combination of ibrutinib and lenalidomide in MDS.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of MDS by World Health Organization (WHO) criteria (including secondary and therapy-related disease) who have failed standard therapy, who are intolerant of prior therapy, or who refuse standard therapy; any prior therapy, including ibrutinib and/or lenalidomide (unless intolerant of one or both of these medications), is permitted

  * Hypomethylating agent failure is defined as disease progression or stable disease as best response to an adequate course of treatment (at least four cycles) with an injectable hypomethylating agent (azacitidine or decitabine)
* International Prognostic Scoring System (IPSS)-revised (R) intermediate, high or very high risk disease
* No specific hematologic parameters for study entry are required; transfusion-dependent patients are eligible and platelet counts should be maintained greater than 10,000/mm^3
* Serum aspartate transaminase (AST) or alanine transaminase (ALT) less than or equal to 3.0 x upper limit of normal (ULN)
* Estimated creatinine clearance greater than or equal to 60 ml/min (Cockcroft-Gault)
* Bilirubin less than or equal to 1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
* Prothrombin time (PT)/international normalized ratio (INR) less than or equal to 1.5 x ULN and partial thromboplastin time (PTT) (activated [a]PTT) less than or equal to 1.5 x ULN
* Karnofsky performance status (KPS) performance status of 60% or greater
* Ability to understand and willingness to sign an informed consent form
* Ability to adhere to the study visit schedule and other protocol requirements
* Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for >= 1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy); or, female subjects of childbearing potential must have a negative serum pregnancy test upon study entry
* Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) during the period of therapy and for 30 days after the last dose of study drug
* Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the Revlimid Risk Evaluation and Mitigation Strategies (REMS) program
* All study participants must be registered into the mandatory Revlimid REMS program, and be willing and able to comply with the requirements of the REMS program
* Eligibility of patients receiving any medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of ibrutinib or ability to adhere to the Revlimid REMS program will be determined following review of their case by the principal investigator

Exclusion Criteria:

* Anticancer therapy including chemotherapy, immunotherapy, radiotherapy, hormonal or any investigational therapy within 14 days or 5 half-lives (whichever is shorter) prior to first dose of study drug; hydroxyurea is permitted up to the day before initiation of study treatment
* Prior allogeneic (allo)-hematopoietic cell transplantation (HCT) less than three months from the time of enrollment
* Acute graft versus host disease (GVHD) or active chronic GVHD greater than grade 1
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration [> 14 days] of > 60 mg/day of prednisone or equivalent) within 28 days of the first dose of study drug
* History of allergy to or intolerance of ibrutinib or lenalidomide
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug
* Recent culture-documented infection requiring systemic intravenous treatment that was completed =< 7 days before the first dose of study drug or any uncontrolled active systemic infection; fever of unknown origin is not an exclusion criterion, as this may be disease-related
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), grade 2 or less, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia
* Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia
* History of stroke or intracranial hemorrhage within 3 months prior to enrollment
* Active infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV) or hepatitis B virus (HBV); subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR positive will be excluded; subjects with HIV must have a CD4 count at or above the institutional lower limit of normal and not taking prohibited CYP3A strong inhibitors
* Major surgery within 4 weeks of first dose of study drug
* Any life-threatening illness, medical condition, or organ system dysfunction, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active autoimmune disorder, or psychiatric illness/social situations that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk
* History of other malignancies, except for malignancy surgically resected (or treated with other modalities) with curative intent, adequately treated in situ carcinoma of the breast or cervix uteri, basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin
* Concomitant use of warfarin or other vitamin K antagonists
* Subjects who received a strong cytochrome P 450 3A (CYP3A) inhibitor within 7 days prior to the first dose of ibrutinib or subjects who require continuous treatment with a strong CYP3A inhibitor
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification
* Lactating or pregnant patients or patients of reproductive potential not willing to use effective methods of contraception and adhere to the Revlimid REMS program
* Participation in clinical trials with other investigational agents not included in this trial throughout the duration of this trial
* Unwilling or unable to participate in all required study evaluations and procedures or unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-11-17 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Up to 28 days
  Data will be reported in tables with descriptive statistics used. Will be assessed by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Effects (CTCAE) version 4.03. Tables will be created to summarize the toxicities and adverse effects by dose, course, organ and severity as well as the study demographics.

SECONDARY OUTCOMES:
Disease free survival | From the time of first documented complete response until relapse or the date of death from any cause, assessed up to 6 months
  Will be summarized with Kaplan-Meier plots.
Disease response | Up to 6 months
  Will be assessed per modified International Working Group (IWG) 2006 response criteria. Response rates and the corresponding 95% confidence intervals will be obtained.
Hematologic normalization rate | Up to 6 months
  Will be assessed as complete remission + partial remission + hematologic improvement.
Overall survival | From the time of first study drug administration until the date of death from any cause, assessed up to 6 months
  Will be summarized with Kaplan-Meier plots.
Progression free survival | From the time of first study drug administration until the date of progression or death from any cause, assessed up to 6 months
  Will be summarized with Kaplan-Meier plots.
Time to response | From the time of first study drug administration to the date of complete remission, partial remission, or hematologic improvement, assessed up to 6 months
  Will be summarized with Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jonas, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States